CLINICAL TRIAL: NCT00018278
Title: Verbal Memory ERPs as Indices of Treatment Response in Alzheimer Disease
Brief Title: Electrophysiologic Measures of Treatment Response in Alzheimer Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AGCG-004-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; Rivastigmine

INTERVENTIONS:
Drug: Aricept
Drug: Exelon
Drug: Nicoderm Patch

SUMMARY:
The main purpose of this study is to determine the electrophysiological effects of cholinergic therapy (cholinesterase inhibitors and transdermal nicotine) in Alzheimer disease. The attempt will be to locate electrophysiological markers and predictors of cognitive and clinical treatment response.

ELIGIBILITY:
Patients diagnosed with mild to moderate probable Alzheimer's disease (mini-mental state exam scores between 15-27), and normal controls (age generally between 60-85). Subjects must either be planning to start daily cholinesterase therapy (e.g. Aricept, Exelon) or willing to try a transdermal nicotine patch for two 8 hour periods.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1998-10; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Vincente Iragui, M.D., Ph.D; Shuanna Morris, Ph.D.
Locations (1):
- Department of Veterans Affairs, San Diego, California, United States